CLINICAL TRIAL: NCT03937999
Title: A Pragmatic Trial of Secondary Prophylaxis With Bezlotoxumab to Prevent C. Difficile Relapse Among Hospitalized Adults Receiving Antibiotics.
Brief Title: Bezlotoxumab as Secondary Prophylaxis for C. Difficile in High-risk Hospitalized Patients Exposed to Antibiotics.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment due to COVID19 , change in practice with standardized use of oral vancomycin prophylaxis
Sponsor: Montefiore Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-10212
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Clostridium Difficile
Keywords: clostridium difficile; diarrhea
MeSH Terms: conditions — Diarrhea | interventions — bezlotoxumab

STUDY DESIGN:
Intervention Model Description: Intervention group compared to concurrent and historical control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bezlotoxumab Arm (Experimental): Single dose of Bezlotoxumab 10mg/kg iv over 60 minutes on Day 0
  Interventions: Drug: Bezlotoxumab
- No Bezlotoxumab (No Intervention): Control group who are eligible as per the inclusion/exclusion criteria to the Bezlotoxumab arm, but not given Bezlotoxumab (Day 0) .

INTERVENTIONS:
Drug: Bezlotoxumab — Injection: 1,000 mg/40 mL (25 mg/mL) solution in a single-dose vial.
  Other Names: Zinplava
  Arms: Bezlotoxumab Arm

SUMMARY:
This study will examine whether the human monoclonal antibody, bezlotoxumab administered AFTER acute Clostridioides difficile (C.diff) has resolved, but during a period of subsequent antibiotic therapy, will eliminate the high risk of C. diff relapse.

DETAILED DESCRIPTION:
Clostridioides difficile (C. diff) is a germ (bacteria) that causes life-threatening diarrhea. It is usually a side-effect of taking antibiotics that affect the normal balance of bacteria in the intestines. When the "good bacteria" in the intestine are killed by antibiotics, the C.diff bacteria begin to grow and produce toxins, causing frequent diarrhea and other symptoms such as abdominal pain or tenderness, loss of appetite, low-grade fever, nausea and vomiting. C. diff can be treated by using special antibiotics, but it tends to come back in about 20% of patients. C-diff is problematic because of frequent relapses after apparent cure. The greatest risk factor for relapse is receipt of subsequent antibiotics, in the hospital, shortly after being treated.

Zinplava™(bezlotoxumab) is an FDA approved human monoclonal antibody designed to prevent the recurrence of C.diff.This is not an antibiotic, as it does not kill C. diff, but is an antibody to C. diff toxins, which stops the damage. When Bezlotoxumab is given during a C. diff infection together with antibiotics to kill C. diff, it decreases the risk that C. diff will come back by about one-half. Bezlotoxumab is approved for use when given during a C. diff infection, but it has not been used to prevent C diff in other situations, such as the one being studied in this research.

ELIGIBILITY:
Inclusion Criteria:

* C diff diagnosed within 90 days
* Receipt of high-risk antibiotics for C diff (e.g. Beta-lactams, carbapenems) in an inpatient setting
* Age 60 years and older

Exclusion Criteria:

* Receipt of current C.diff active antibiotics (oral vancomycin, fidaxomycin, metronidazole, tigecycline/ doxycycline, nitazoxanide, rifamycin) within 72hrs.
* Not Expected to survive 8 weeks
* Prior or planned fecal microbiota transplant or Bezlotoxumab use
* Congestive heart failure (a potential risk of Bezlotoxumab)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Riska, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bezlotoxumab Arm | No Bezlotoxumab
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled in the study (control group). Study terminated early due to lack of enrollment
Groups:
- No Bezlotoxumab: Control group who are eligible as per the inclusion/exclusion criteria to the Bezlotoxumab arm, but not given Bezlotoxumab (Day 0).
- Total: Total of all reporting groups
Arm/Group | Bezlotoxumab Arm | No Bezlotoxumab | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of C.Difficile Infection
Time Frame: within 4 weeks
Population: Only 1 participant was enrolled in the study (into the 'No Bezlotoxumab' control group). No statistical analysis was conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Bezlotoxumab Arm | No Bezlotoxumab
Number analyzed (Participants) | 0 | 1
Participants |  | 0

2. Secondary Outcome: Recurrence of C.Difficile Infection
Time Frame: within 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bezlotoxumab Arm | No Bezlotoxumab
Number analyzed (Participants) | 0 | 1
Participants |  | 0

3. Secondary Outcome: Rate of Deaths
Time Frame: within 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bezlotoxumab Arm | No Bezlotoxumab
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 0

4. Secondary Outcome: Relapse of C. Difficile by 8 Weeks
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bezlotoxumab Arm | No Bezlotoxumab
Number analyzed (Participants) | 0 | 1
Participants |  | 1

ADVERSE EVENTS:
Time Frame: Participants queried at 1 day, 4 weeks, and 8 weeks
Description: No participants were enrolled into the treatment into the Bezlotoxumab Arm of the study.
Arm/Group | Bezlotoxumab Arm | No Bezlotoxumab
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03937999/Prot_SAP_000.pdf